CLINICAL TRIAL: NCT05532111
Title: Efficacy and Safety of Rituximab Combined With Tacrolimus in the Treatment of Intermediate-to-high Risk Primary Membranous Nephropathy: A Randomized Clinical Trial
Brief Title: Efficacy and Safety of the Treatment of Primary Membranous Nephropathy: A Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2021-0149
Record Dates: First submitted 2022-09-01; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Efficacy and Safety
Keywords: Rituximab; Tacrolimus; Primary Membranous Nephropathy
MeSH Terms: interventions — Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- RT-R Group (Experimental): Rituximab combined with tacrolimus induction + rituximab maintenance
  Interventions: Drug: Rituximab combined with tacrolimus induction + rituximab maintenance
- RT-T Group (Experimental): Rituximab combined with tacrolimus induction + tacrolimus maintenance
  Interventions: Drug: Rituximab combined with tacrolimus induction + tacrolimus maintenance
- PC-C Group (Experimental): Glucocorticoid combined with cyclophosphamide induction + maintenance
  Interventions: Drug: Glucocorticoid combined with cyclophosphamide induction + maintenance

INTERVENTIONS:
Drug: Rituximab combined with tacrolimus induction + rituximab maintenance — RT-R group: Rituximab 1 g/time, once in 15 days, × 2 times, combined with tacrolimus, the initial dose is 0.05-0.1 mg/kg/d, 2 times at an interval of 12 hours, orally. Adjust the dose according to the blood concentration (maintain the blood concentration C0 4-8ng/ml). At the end of 24 weeks, tacrolimus was stopped, and rituximab was given 1 g/time × 1 time.
  Arms: RT-R Group
Drug: Rituximab combined with tacrolimus induction + tacrolimus maintenance — RT-T group: Rituximab 1 g/time, once in 15 days, × 2 times, combined with tacrolimus, the initial dose is 0.05-0.1 mg/kg/d, 2 times at an interval of 12 hours, orally. Adjust the dose according to the blood concentration (maintain the blood concentration C0 4-8ng/ml).
  Arms: RT-T Group
Drug: Glucocorticoid combined with cyclophosphamide induction + maintenance — PC-C group: The initial dose of prednisone/prednisolone was 0.5-1 mg/kg/d (the maximum dose was 70 mg/d), and the dose was gradually reduced after 4-8 weeks, and then stopped within 6-9 months. Cyclophosphamide 750mg/m2 (adjusted according to eGFR and other conditions), once a month, intravenous pulse therapy. CTX maintenance therapy.
  Arms: PC-C Group

SUMMARY:
1. Main purpose:

   To evaluate the efficacy and safety of rituximab combined with tacrolimus in the treatment of intermediate and high-risk primary membranous nephropathy
2. Secondary research purposes:

   To describe the survival of patients with intermediate and high-risk primary membranous nephropathy treated with rituximab combined with tacrolimus; To describe renal survival in patients with intermediate and high-risk primary membranous nephropathy treated with rituximab combined with tacrolimus;
3. Exploratory research purposes:

Feasibility of glucocorticoids-free therapy (rituximab combined with tacrolimus) in the treatment of intermediate and high-risk primary membranous nephropathy

DETAILED DESCRIPTION:
Membranous nephropathy (MN) is the leading cause of primary nephrotic syndrome in adults, with a peak incidence in middle-aged and elderly patients. The typical pathological features are: thickening of the basement membrane, deposition of immunofluorescent IgG with or without C3 along the basement membrane, and deposition of epithelial electron-dense deposits. It is divided into primary MN (Primary membranous nephropathy, PMN) and secondary MN (which can be secondary to connective tissue diseases, infections, malignant tumors, drugs/toxicants, etc.). Clinically, it usually presents with massive proteinuria and edema, and some patients gradually progress to end stage renal disease (ESRD).

In recent years, the prevalence of PMN in China has increased year by year. It has been reported that the proportion of MN in primary glomerular diseases in renal biopsy increased from 10.4% in 2003-2006 to 24.1% in 2011-2014 [1], and some trend of youth.

For a long time, the treatment of PMN has mainly used glucocorticoids combined with alkylating agents or calcineurin inhibitors (CNIs). With the continuous exploration and in-depth understanding of the pathogenesis of MN, it has been developed to the molecular level. The KDIGO 2021 Glomerular Disease Management Guidelines are being published [2] Compared with the 2012 KDIGO Glomerular Disease Management Guidelines, the diagnosis and treatment of MN has undergone major changes (Figure 1). Due to the toxicity of alkylating agents and the long-term nephrotoxicity of CNIs, as well as their high risk of relapse when used as monotherapy (with or without prednisone), anti-CD20 biotherapeutics (especially Rituximab, RTX)) is gaining popularity as first-line therapy.

Both international and domestic guidelines recommend that moderate and severe MN require immunosuppressive therapy. RTX is an anti-CD20 monoclonal antibody, which can block the generation of B cells, differentiate into plasma cells, reduce the production of antibodies (such as PLA2R), and avoid processes such as glomerular basement membrane damage. TAC is a calcineurin inhibitor that has been used in PMN for many years. It mainly acts through various mechanisms such as immune regulation and stabilization of the pod cytoskeleton. Two-drug sequential therapy can work from multiple mechanisms, potentially achieving better and faster therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* gender is not limited；
* Age 18-75；
* Kidney biopsy pathology suggests primary membranous nephropathy;
* Serological or histological PLA2R positive;
* 24-hour urine protein quantification ≥3.5g/d and serum albumin <30g/L;
* Glomerular filtration rate [eGRF (CKD-EPI formula)] ≥ 45ml/min/1.73m2;

Exclusion Criteria:

* Secondary membranous nephropathy (tumor-related, lupus-related, hepatitis B-related, infection-related, drug-related, etc.);
* Renal biopsy pathology showed severe tubulointerstitial lesions;
* Severe infection, severe cardiac insufficiency, severe hepatic insufficiency, gastrointestinal bleeding, ketoacidosis and other life-threatening complications within one month;
* Glucocorticoids and/or immunosuppressive therapy (cyclophosphamide, MMF, tacrolimus) within 3 months;
* Have a history of kidney transplantation;
* Breastfeeding or pregnant women;
* Patients with mental disorders or unable to cooperate ;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
24-hour urine protein quantification | 48 weeks
  1. Remission: decreased proteinuria. Complete remission (CR): 24HUTP<0.3g/L Partial remission (PR): 24HUTP decreased by >50% and >0.3g/L from baseline
  2. Invalid: no decrease in proteinuria compared with baseline.
  3. Recurrence: increased proteinuria (24-hour urine protein quantification ≥3.5g/d) , recurred after reaching CR or PR.
serum albumin | 48 weeks
  1. Remission: serum albumin>30g/L
  2. Invalid: serum albumin <30g/L
  3. Recurrence: decreased serum albumin, <30g/L, recurred after reaching CR or PR.